CLINICAL TRIAL: NCT05267002
Title: One Week Versus Two Week Removal of Nylon Cutaneous Sutures for Linear Layered Closures on the Face: a Randomized Evaluator-blinded Prospective Split-scar Trial
Brief Title: Comparing 1 Week Versus 2 Week Cutaneous Suture Removal
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: DermSurgery Associates (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 9728
Record Dates: First submitted 2022-02-24; First posted 2022-03-04 (Actual); Last update posted 2022-03-04 (Actual); Status verified 2022-02

CONDITIONS: Suture; Complications, Mechanical; Scar; Surgery
MeSH Terms: conditions — Cicatrix

STUDY DESIGN:
Intervention Model Description: Split Scar Study
Who Masked: Outcomes Assessor
Masking Description: The primary outcome will be the Scar Cosmesis Assessment and Rating scale (SCAR) score, with photographic assessment by three blinded fellowship-trained board-certified Mohs surgeons who were not involved with the original surgery or wound repair.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Suture removal at 1 week (Experimental): Cutaneous nylon suture removal of half of the split-scar at one week.
  Interventions: Procedure: Suture removal timing
- Suture removal at 2 weeks (Experimental): Cutaneous nylon suture removal of half of the split-scar at two weeks.
  Interventions: Procedure: Suture removal timing

INTERVENTIONS:
Procedure: Suture removal timing — Cutaneous nylon suture removal of each half of the split-scar at one and two weeks.

SUMMARY:
Our goal is to compare the difference in surgical outcomes and patient satisfaction for surgical scars on the face between suture removal at 1 week versus 2 weeks.

There is variation in the timing at which Mohs surgeons remove sutures on the face. Some prefer 1 week, and others prefer 2 weeks. This has not been formally studied. It is possible the outcomes are the same between both groups, or that one has a better cosmetic outcome than the other.

Your skin cancer will be removed as usual. After this, your wound will be sutured in the usual fashion, except the top sutures will be divided into two separate halves. You will return at 1 week for one half of the top sutures to be removed, and at 2 weeks for the other half to be removed. Which half is removed first will be determined at random at your 1 week visit. At two months, you will return for standardized photographs which will be used by physicians to rate the cosmetic outcomes of the wound halves based on a standardized scale. Most likely, there will be no difference between the wound halves at 2 months and the study is complete. There is a small chance that there will be a cosmetic difference seen at 2 months, in which case you will return at 1 year for repeat standardized photographs and ratings. All data and photographs will be kept secure and any identifying information will be destroyed at the end of the study.

DETAILED DESCRIPTION:
This is an investigator initiated, single-center, prospective, randomized, evaluator-blinded split-scar study. Subjects will be recruited at the time of repair for Mohs surgery or excision based on the inclusion criteria above. Procedures will be performed by fellowship trained Mohs surgeons or fellows in training. The same surgeon will close the entire wound. At the time of wound closure, the wound will be divided into two equal halves. Subcutaneous 4-0 or 5-0 polyglecaprone sutures will be used to fully approximate the wound edges. Subcutaneous sutures will begin with one subcutaneous suture immediately in the center of the wound, followed by symmetrical subcutaneous sutures on both sides of the defect until the wound edges are approximated.

Once the wound edges are approximated, 5-0 nylon sutures will be used to align the epidermal edges in a running fashion, with sutures spaced 3-5mm apart and 2-3 mm from the wound edge. Suturing will begin at the wound poles and run towards the center. The running nylon sutures will be tied off separately for each wound half, which will facilitate suture removal in 1 or 2 weeks. Order of suturing the halves will be at the preference of the surgeon, as randomization will take place later at suture removal. The entire wound will then be dressed with a bandage, which will be left on 24 hours, at which point they may wash the site and change the bandage daily.

The patient will next present at 1 week (7 days) for randomization and suture removal of one half. The half that is either superior or on the patient's right will be labeled "A," and the other half will be labeled "B". This labeling will be photographed into the patient's electronic medical record and will be kept consistent for the remainder of the study. The patient will then be randomized using a random number generator (random.org), generating a number 1 or 2. If randomization yields a 1, then half A is removed first. If randomization yields a 2, then half B is removed first. The patient will return again at 2 weeks for removal of the second half of the nylon sutures.

At two months, patients will have standardized wound photographs taken: the wound will be re-labeled with "A" or "B" as it was at the time of suture removal. A Nikon SLR camera with 105mm macro lens, Wireless speedlight mounted on a ring, aperture F11, shutter 1/250 second, and Iso 64 will be consistent for all photographs. A standard grey background will be used, and the photograph will be taken at 90 degrees to the wound with the full face filling the frame.

The primary outcome will be the Scar Cosmesis Assessment and Rating scale (SCAR) score, with photographic assessment by three blinded fellowship-trained board-certified Mohs surgeons who were not involved with the original surgery or wound repair. There will be a preliminary statistical analysis, and if there is no difference between groups at 2-months, then the study will be ended (prior research has shown that if there is no difference at interim follow up, then the probability of difference at 1-year follow up is low enough as to not justify additional office visits for the patient). If there is a statistical difference seen at 2-months, then the study will continue through a 12-month visit, at which point repeat clinical photographs will be taken and evaluated as above.

ELIGIBILITY:
Inclusion Criteria i. Adult patients >18 years ii. Undergoing Mohs surgery or excision with layered repair

1. intermediate or complex layered closures measuring 2.6-7.5 cm on the face (including the forehead, temples, nose, cheeks, chin)
2. Wound edges must be able to be approximated with subcutaneous sutures. iii. Ability to follow up at 1 week, 2 weeks, 2 months, and 1 year iv. Participants able to be enrolled at time of wound repair.

Exclusion criteria i. Facial defects involving the eyelid, mucosal lip, and ear ii. Pregnant or breastfeeding women iii. Children <18 years iv. Inability to comprehend English v. Inability to consent vi. Incarceration

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2022-02-24 (Actual); Primary Completion 2023-05-24 (Estimated); Study Completion 2023-05-24 (Estimated)

PRIMARY OUTCOMES:
Scar Cosmesis Assessment and Rating scale (SCAR) score | 2months (and possibly one year, see protocol)
  1. Scar Cosmesis Assessment and Rating scale (SCAR), rated by three blinded observers based on digital photographs, with each half of the scar scored separately. This is a 0-13 rating with 0 representing the best possible scar.

SECONDARY OUTCOMES:
pain level with suture removal | measured at 1 and 2 weeks after suture removal
  0-10 scale
difficulty of suture removal | measured at 1 and 2 weeks
  provider ranked difficulty of suture removal (easy, moderate or difficult)
Patient scar satisfaction | At 2 months
  patients will rate "how satisfied are you with the scar" on a 0-10 point scale (10= most satisfied) on each half of the wound
Patient preference for 1 vs 2 week suture removal. | Asked at 2 months
  At the 2-month visit patients will be asked whether they prefer 1 week or 2 week suture removal (answer choices will be 1 week/2 week/no preference). If they have a preference, an open-ended question as to why will be asked.
Presence of suture tracks | 2 months
  Whether or not suture track marks were present at 2 months.
Rates of complications | 2 months
  Rates of complications (dehiscence, infection, hematoma, deep suture reaction) on each half of the wound.

CONTACTS AND LOCATIONS:
Overall Officials: Leonard H Goldberg, MD, Study Director — DermSurgery Associates
Locations (1):
- DermSurgery Associates, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Eisen DB, Zhuang AR, Hasan A, Sharon VR, Bang H, Crispin MK. 5-0 Polypropylene versus 5-0 fast absorbing plain gut for cutaneous wound closure: a randomized evaluator blind trial. Arch Dermatol Res. 2020 Apr;312(3):179-185. doi: 10.1007/s00403-019-02009-5. Epub 2019 Nov 13. PMID 31724097
- [Background] Yag-Howard C. Sutures, needles, and tissue adhesives: a review for dermatologic surgery. Dermatol Surg. 2014 Sep;40 Suppl 9:S3-S15. doi: 10.1097/01.DSS.0000452738.23278.2d. PMID 25158874
- [Background] Gal P, Toporcer T, Vidinsky B, Hudak R, Zivcak J, Sabo J. Simple interrupted percutaneous suture versus intradermal running suture for wound tensile strength measurement in rats: a technical note. Eur Surg Res. 2009;43(1):61-5. doi: 10.1159/000219214. Epub 2009 May 19. PMID 19451720
- [Background] Joo JS, Zhuang AR, Tchanque-Fossuo C, Tartar D, Armstrong AW, King TH, Sivamani RK, Eisen DB. Dermal suture only versus layered closure: A randomized, split wound comparative effectiveness trial. J Am Acad Dermatol. 2019 Dec;81(6):1346-1352. doi: 10.1016/j.jaad.2019.08.040. Epub 2019 Aug 21. PMID 31442535
- [Background] Kantor J. Reliability and Photographic Equivalency of the Scar Cosmesis Assessment and Rating (SCAR) Scale, an Outcome Measure for Postoperative Scars. JAMA Dermatol. 2017 Jan 1;153(1):55-60. doi: 10.1001/jamadermatol.2016.3757. PMID 27806156